CLINICAL TRIAL: NCT00218777
Title: Behavior Therapy for Children With Chronic Tic Disorders
Brief Title: Cognitive Behavior Therapy and Habit Reversal Training for the Treatment of Chronic Tic Disorders in Children
Acronym: CBIT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tourette Association of America (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, John Piacentini, Chair, TSA Behavioral Sciences Consortium; Director, UCLA Child OCD, Anxiety and Tic Disorders Program, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH070802 (NIH); R01MH070802 (NIH); DSIR 84-CTS
Record Dates: First submitted 2005-09-21; First posted 2005-09-22 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Tourette Syndrome; Tic Disorders
Keywords: Chronic tic disorder; Motor tics; Vocal tics
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders; Tics

INTERVENTIONS:
Behavioral: Comprehensive Behavioral Intervention for Tics

SUMMARY:
This study will determine the effectiveness of cognitive behavior therapy (CBT) with habit reversal training (HRT) in treating chronic tic disorders (CTDs) in children and adolescents.

DETAILED DESCRIPTION:
CTDs and Tourette syndrome are neurobehavioral disorders that are characterized by a persistent pattern of motor and vocal tics. Tics are intermittent movements or sounds that occur repeatedly. They can be either brief, rapid, and darting movements or more purposeful movements, such as repetitively locking and unlocking a door. Vocal tics can be simple, as in sniffing or grunting, or more complex, such as complete words or phrases. Tic disorders can cause considerable distress in affected children, and can lead to social and academic impairment. If left untreated, CTDs can last into adulthood. The standard treatment for suppressing CTDs is medication; dopamine-blocking drugs are used most commonly. These medications, however, are associated with a range of adverse effects that can result in poor treatment compliance and premature treatment termination. Recent research suggests that HRT may be an effective, lower risk treatment for CTDs. HRT is a behavioral treatment based on increasing awareness of one's behaviors and replacing unwanted behaviors with less bothersome ones. This study will determine the effectiveness of CBT with HRT in treating CTDs in children and adolescents.

Participants in this double blind study will be randomly assigned to receive either CBT plus HRT or standard care, which will consist of psychoeducation and supportive therapy. All participants will partake in 8 sessions of their assigned therapy over the course of 10 weeks. After the initial 10 weeks, those who responded to treatment will report back to the study site for 3 monthly booster sessions. Changes in tic severity, effects of the therapies on overall functioning and quality of life, and possible predictors of treatment outcome will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV diagnostic criteria for chronic tic disorder (chronic motor or vocal tic disorder or Tourette syndrome)
* Score of at least 3 on the Clinical Global Impressions Severity Scale
* Score of at least 14 on the Yale Global Tic Severity Scale (YGTSS) or at least 10 for individuals with motor tics only
* Unmedicated or currently on a stable medication treatment for tics, obsessive compulsive disorder (OCD), ADHD, anxiety, and/or depressive disorder for at least 6 weeks, with no planned changes for the duration of study participation
* Child speaks English

Exclusion Criteria:

* Score greater than 30 on the YGTSS
* IQ less than 80 on the Wechsler Abbreviated Scale of Intelligence (WASI)
* Meets DSM-IV criteria for substance abuse or dependence within the 3 months prior to study entry
* Meets DSM-IV criteria for conduct disorder within the 3 months prior to study entry
* Lifetime DSM-IV diagnosis of pervasive developmental disorder, mania, or psychotic disorder
* Any serious psychiatric, psychosocial, or neurological condition (i.e., OCD, ADHD, major depressive disorder, anxiety, severe aggression, or family discord) requiring immediate treatment other than what is provided in the current study (i.e., medication, school intervention, or family therapy)
* Previous treatment with four or more sessions of HRT for tics

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2004-12; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Reduction in tic severity | 10-22 weeks
Reduction in tic-related impairment and distress (measured at Week 10) | measured at week 10

SECONDARY OUTCOMES:
Tic severity and associated impairment and distress (measured at Week 36 follow-up) | measured at week 36 follow-up
Changes in neurocognitive function (measured at Week 10) | measured at week 10

CONTACTS AND LOCATIONS:
Overall Officials: John Piacentini, PhD, Principal Investigator — University of California at Los Angeles
Locations (3):
- United States (3):
  - UCLA Child OCD, Anxiety, and Tic Disorders Program, Los Angeles, California
  - Johns Hopkins University, Baltimore, Maryland
  - University of Wisconsin-Milwaukee, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Houghton DC, Capriotti MR, Scahill LD, Wilhelm S, Peterson AL, Walkup JT, Piacentini J, Woods DW. Investigating Habituation to Premonitory Urges in Behavior Therapy for Tic Disorders. Behav Ther. 2017 Nov;48(6):834-846. doi: 10.1016/j.beth.2017.08.004. Epub 2017 Aug 10. PMID 29029679
- [Derived] Sukhodolsky DG, Woods DW, Piacentini J, Wilhelm S, Peterson AL, Katsovich L, Dziura J, Walkup JT, Scahill L. Moderators and predictors of response to behavior therapy for tics in Tourette syndrome. Neurology. 2017 Mar 14;88(11):1029-1036. doi: 10.1212/WNL.0000000000003710. Epub 2017 Feb 15. PMID 28202705
- [Derived] Peterson AL, McGuire JF, Wilhelm S, Piacentini J, Woods DW, Walkup JT, Hatch JP, Villarreal R, Scahill L. An Empirical Examination of Symptom Substitution Associated With Behavior Therapy for Tourette's Disorder. Behav Ther. 2016 Jan;47(1):29-41. doi: 10.1016/j.beth.2015.09.001. Epub 2015 Sep 11. PMID 26763495
- [Derived] McGuire JF, Piacentini J, Scahill L, Woods DW, Villarreal R, Wilhelm S, Walkup JT, Peterson AL. Bothersome tics in patients with chronic tic disorders: Characteristics and individualized treatment response to behavior therapy. Behav Res Ther. 2015 Jul;70:56-63. doi: 10.1016/j.brat.2015.05.006. Epub 2015 May 12. PMID 25988365
- [Derived] McGuire JF, Nyirabahizi E, Kircanski K, Piacentini J, Peterson AL, Woods DW, Wilhelm S, Walkup JT, Scahill L. A cluster analysis of tic symptoms in children and adults with Tourette syndrome: clinical correlates and treatment outcome. Psychiatry Res. 2013 Dec 30;210(3):1198-204. doi: 10.1016/j.psychres.2013.09.021. Epub 2013 Sep 27. PMID 24144615
- [Derived] Jeon S, Walkup JT, Woods DW, Peterson A, Piacentini J, Wilhelm S, Katsovich L, McGuire JF, Dziura J, Scahill L. Detecting a clinically meaningful change in tic severity in Tourette syndrome: a comparison of three methods. Contemp Clin Trials. 2013 Nov;36(2):414-20. doi: 10.1016/j.cct.2013.08.012. Epub 2013 Aug 31. PMID 24001701
- [Derived] Woods DW, Piacentini JC, Scahill L, Peterson AL, Wilhelm S, Chang S, Deckersbach T, McGuire J, Specht M, Conelea CA, Rozenman M, Dzuria J, Liu H, Levi-Pearl S, Walkup JT. Behavior therapy for tics in children: acute and long-term effects on psychiatric and psychosocial functioning. J Child Neurol. 2011 Jul;26(7):858-65. doi: 10.1177/0883073810397046. Epub 2011 May 9. PMID 21555779
- [Derived] Piacentini J, Woods DW, Scahill L, Wilhelm S, Peterson AL, Chang S, Ginsburg GS, Deckersbach T, Dziura J, Levi-Pearl S, Walkup JT. Behavior therapy for children with Tourette disorder: a randomized controlled trial. JAMA. 2010 May 19;303(19):1929-37. doi: 10.1001/jama.2010.607. PMID 20483969
- See also: Click here for the Tourette Syndrome Association, Inc. website — http://www.tsa-usa.org/